CLINICAL TRIAL: NCT02817789
Title: Safety Profile Evaluation of TICagrelor Alone Compared to a Combination of Lysine Acetylsalicylate-Clopidogrel in the Context of Transcatheter Aortic Valve Implantation (TAVI)
Acronym: TICTAVI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2014/24
Record Dates: First submitted 2016-04-29; First posted 2016-06-29 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; Antiplatelet agent; Ticagrelor; Cerebrovascular events
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard group (Active Comparator): 154 patients
  Interventions: Drug: Combination lysine acetylsalicylate - clopidogrel
- Ticagrelor group (Experimental): 154 patients
  Interventions: Drug: Ticagrelor alone

INTERVENTIONS:
Drug: Ticagrelor alone — 180 mg loading dose before intervention and 90 mg twice daily during 30 days after the procedure
  Arms: Ticagrelor group
Drug: Combination lysine acetylsalicylate - clopidogrel — 75 mg before and 75 mg daily after the procedure of lysine acetylsalicylate and 300mg loading dose before and 75 mg of clopidogrel daily after the procedure
  Arms: Standard group

SUMMARY:
Transcatheter Aortic Valve Implantation (TAVI) is now the method of choice to treat aortic stenosis in old and frail patients. Antiplatelet therapy must be associated for the procedure and during few weeks after implantation in the aim to minimize cerebral embolization. But for now, the best antiplatelet regimen has to be determined. In this context, investigators want to evaluate the safety of use of ticagrelor alone versus standardized therapy which involves lysine acetylsalicylate and clopidogrel. In this study, we will randomly compare 154 patients in each group in terms of early safety (30 days) after the procedure.

DETAILED DESCRIPTION:
In spite of the use of the combination of lysine acetylsalicylate and clopidogrel during and after the procedure of TAVI, rates of stroke remains high, between 4 and 10% regarding the studies and registries. None of the therapeutics have regulatory authorisation for this indication. On the other hand, the rates of bleeding events are also high in this old and frail population. That is why, considering its pharmacological specificity, investigators hypothesize that ticagrelor, used alone, could be non-inferior on safety criteria than the combination of lysine acetylsalicylate and clopidogrel. Our study want to evaluate the safety profile of Ticagrelor alone (180 mg loading dose before intervention and 90 mg twice daily during 30 days after the procedure) compared to the standardized treatment combining lysine acetylsalicylate (75 mg before and 75 mg daily after the procedure) and clopidogrel (300mg loading dose before and 75 mg daily after the procedure). Patients will be followed during one month. Then they will be all placed under the usual antiplatelet treatment (clopidogrel and lysine acetylsalicylate for two additional months and then lysine acetylsalicylate alone lifelong).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female or male aged > 18 years
* Patient eligible for TAVI as recommended by French health care system authority (HAS)

Exclusion Criteria:

* Allergy, hypersensitivity, or contraindication to lysine acetylsalicylate, clopidogrel, ticagrelor, any anticoagulation or magnetic resonance imaging (MRI) or CT-scanner contrast agents
* Use of Cytochrome P3a (CYP3a) inhibitor
* Need for chronic anticoagulation
* Previous percutaneous coronary intervention or acute coronary syndrome requiring dual antiplatelet therapy
* Previous cardiac surgery for valve replacement
* Prior stroke, transient ischemic attack (TIA) or known carotid stenosis > 70%
* Active pathological bleeding or gastric ulcer < 3month
* Known thrombocytopenia, anemia or any coagulopathy
* Severe kidney or hepatic impairment
* Hemodynamic instability
* Refusal of Transfusion
* Significant mental impairment
* Inability to give informed consent or comply with study related procedures or high likelihood of being unavailable for follow-up
* Pregnant or breastfeeding women
* Women of childbearing potential without effective contraception (oestroprogestative, intrauterine devices)
* Participant in another investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Number of patient presenting at least one event of the Valve Academic Research Consortium-2 (VARC2) composite endpoint | Day 30
  VARC2 composite endpoint :
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening or disabling bleeding
  * Acute kidney injury - Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure
Number of patient died | Day 30
Number of patient presenting stroke or Transient Ischemic Attack (TIA) | Day 30
  Diagnostic criteria: Acute episode of a focal or global neurological deficit with at least one of the following: change in the level of consciousness, hemiplegia, hemiparesis, numbness, or sensory loss affecting one side of the body, dysphasia or aphasia, hemianopia, amaurosis fugax, or other neurological signs or symptoms consistent with stroke Stroke: duration of a focal or global neurological deficit >24 h; OR <24 h if available neuroimaging documents a new haemorrhage or infarct; OR the neurological deficit results in death TIA: duration of a focal or global neurological deficit <24 h, any variable neuroimaging does not demonstrate a new hemorrhage or infarct
Number of patient presenting life-threatening bleeding | Day 30
  Life-threatening bleeding:
  Fatal bleeding OR Bleeding in a critical organ, such as intracranial, intraspinal, intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome OR Bleeding causing hypovolaemic shock or severe hypotension requiring vasopressors or surgery OR Overt source of bleeding with drop in haemoglobin >5 g/dL or whole blood or packed red blood cells (RBCs) transfusion >4 units
Number of patients presenting post-TAVI acute kidney failure stage 2 or 3 as assessed by VARC2 | Day 30
Number of patients presenting angiographic or echographic evidence of a new, partial or complete, obstruction of a coronary ostium, either by the valve prosthesis itself, the native leaflets, calcifications, or dissection | Day 30
Number of patients presenting major vascular complications | Day 30
Number of patients requiring a new procedure like Balloon Aortic valvuloplasty (BAV), new procedure of TAVI or Surgical aortic valve replacement (SAVR) | Day 30

SECONDARY OUTCOMES:
Number of patients presenting at least one conduction disturbance or arrhythmias | Day 30
Number of patients presenting at least one other TAVI related complication | Day 30
Number of patients presenting at least one bleeding event (life-threatening, major or minor) | Day 30
Number of patients with good biological efficiency of the antiplatelet therapy assessed by VerifyNow (VN) | Day 30
Number of patients with new cerebral event assessed by brain Magnetic Resonance Imaging (MRI) | Day 5
Number of high-intensity transient signals (HITS) assessed by transcranial Doppler | Day 1
Assessment of neurological status by the score of Mini Mental State Examination (MMSE) | At baseline and day 30
Assessment of neurological status by the Dubois's 5 words test | At baseline and day 30
Assessment of neurological status by the Geriatric Depression Scale (GDS) | At baseline and day 30
Assessment of neurological status by the basic Activities of Daily Living (ADL) questionnaire | At baseline and day 30
Assessment of neurological status by the Instrumental Activities of Daily Life (IADL) questionnaire | At baseline and day 30
Assessment of neurological status by the Short Form Health Survey (SF-12) questionnaire | At baseline and day 30

CONTACTS AND LOCATIONS:
Overall Officials: Lionel LEROUX, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHRU de Lille, Lille
  - APHM, Marseille
  - CHRU de Nîmes, Nîmes
  - APHP, Paris
  - CHU de Bordeaux, Pessac